CLINICAL TRIAL: NCT02426567
Title: An Exploratory Study on the Impact of a Food-based Restrictive Diet (Crohn's Disease-TReatment-with EATing/CD-TREAT Diet) and Liquid Exclusive Enteral Nutrition (EEN) on Healthy Gut Microbiota Composition and Metabolic Activity
Brief Title: The Impact of "Crohn's Disease-TReatment-with-EATing" Diet and Exclusive Enteral Nutrition on Healthy Gut Bacteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Konstantinos Gerasimidis, Lecturer in Clinical Nutrition, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200130161
Record Dates: First submitted 2015-04-17; First posted 2015-04-27 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Crohn's Disease; Dietary Modification
Keywords: Crohn's Disease; Exclusive Enteral Nutrition; Dietary Treatment; Gut microbiota
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Adult Participants A (Experimental): Participants who will get two interventional diets, for 7 days each, but allocated to start with Exclusive Enteral Nutrition (EEN)
  Interventions: Other: Exclusive Enteral Nutrition (EEN); Other: Crohn's Disease TReatment-with-EATing diet (CD-TREAT diet)
- Healthy Adult Participants B (Experimental): Participants who will get two interventional diets, for 7 days each, but allocated to start with Crohn's Disease TReatment-with-EATing diet (CD-TREAT diet)
  Interventions: Other: Exclusive Enteral Nutrition (EEN); Other: Crohn's Disease TReatment-with-EATing diet (CD-TREAT diet)

INTERVENTIONS:
Other: Exclusive Enteral Nutrition (EEN) — One week course of an isocaloric exclusive milk-based diet
Other: Crohn's Disease TReatment-with-EATing diet (CD-TREAT diet) — One week course of an isocaloric, exclusion food-based diet

SUMMARY:
Current evidence suggests that the gut microbiota and dietary influences are as important as genetics in the aetiology of Crohn's disease (CD). We have recently shown that disease improvement, following treatment with Exclusive Enteral Nutrition (EEN), coincided with changes in the gut microbiota.

The main purposes of this study are: a) to explore whether the gut microbiota changes we observed in this previous study in children with CD during EEN are disease specific or not, and b) to develop a novel food-based diet (Crohn's Disease TReatment-with-EATing/CD-TREAT diet) which will induce changes to the metabolic activity and bacterial composition of the gut microbiota of healthy people, similar to those seen on EEN, the first-line treatment for active paediatric CD.

This study will produce high quality scientific evidence to move the CD-TREAT diet towards a preliminary clinical trial in patients with CD which is currently inappropriate and unethical to carry out in people with active CD undertaking contemporary medical treatment.

DETAILED DESCRIPTION:
This study is a randomised, cross-over, dietary intervention trial. Healthy adult (>18 y) participants from the community will be recruited by means of an advertisement leaflet and word of mouth. Eligible participants will be enrolled in the study. We will thank those subjects who have expressed an interest about the study but are not suitable to participate and we will explain to them why they need to be excluded. Those who are eligible and willing to participate will be asked to undertake two different experimental diets, for seven days each:

1. Exclusive Enteral Nutrition (EEN) which is the exclusive consumption of a milk-based proprietary dietary supplement (Modulen®, Nestle). This is a liquid based diet used for the management of children with active CD. Although this diet is used primary for clinical reasons it is food based and does not contain any drugs or non-food based pharmaceutical ingredients. It is available online and without prescription from pharmacist.
2. Crohn's Disease TReatment-with-EATing diet (CD-TREAT diet), an elimination customized diet which will consist of ordinary food and which will resemble the food/nutrient composition of EEN (e.g. fibre content, fatty acid composition) and considering evidence that implicates certain nutrients, and food ingredients (e.g. meat, sugar) in the aetiology and risk of relapse of CD. Diet will be created using the food group exchange methodology and will be analysed using Windiets® 2010.

Both diets will have the same energy content and will be isocaloric aiming to keep participants' weight stable during the study period. Their energy content will be tailored to participants' total energy expenditure and physical activity level calculated by the WHO set of equations. The order of the diets will be randomly allocated using an MS Excel command. In order to minimize fatigue with the diet but also to ensure that we will be able to detect changes in gut microbiota, experimental diets will be given for 7 days. This is based on recent evidence suggesting that dietary changes for 5 days induce reproducible alterations in gut microbiota composition and metabolism. Prior to the first diet intervention, participants will also record their dietary intake using a 7-day estimated food diary. Between the two interventions the participants will have to eat their habitual diet for two weeks and this will be a wash out period which aims to drive the gut microbiota back to baseline levels. The week prior to the initiation of the second intervention the participants will be asked to keep the same dietary pattern as they had the week prior to the first trial.

Detailed methods:

Preliminary Health Check: Participants will undertake a short health questionnaire including basic health information, age or any medication on the day of recruitment.

Anthropometry: All participants will have height and weight measured at baseline and only weight measured in each sample collection timepoint.

Diet compliance: Over the course of the two experimental diets we will monitor compliance by asking participants to complete a questionnaire. The questionnaire will ask if they felt the need to supplement the diets at any time with other foods or drinks. An interval call 2 days after each diet's initiation will also be used to increase participants' motivation and compliance on the diets.

Sample collection & analysis: Fresh faecal and urine samples will be collected before and after each dietary intervention (4 times in total) to assess and compare the impact of these diets on gut microbiota composition and metabolic activity.

Lab Assays:

1. The gut bacterial diversity and composition from stool samples will be measured using molecular techniques such as quantitative polymerase chain reaction (PCR) from bacterial ribosomal DNA and next generation sequencing (metagenomics).
2. A large number of different products from bacterial metabolism, such as short chain fatty acids, sulphide, and ammonia will be measured using a range of techniques including gas chromatography and gas chromatography mass spectrometry (GCMS)(metabolomics). Faecal pH, a marker of bacterial fermentation, will also be measured.

Power calculation: Fresh faecal and urine samples will be collected from 38 healthy participants at 4 time points. Based on our previous in vivo work in children with CD this would give us a power of 80% (p=0.05) to detect a mean concentration difference of 1.0 log (SD:1.5) in Faecalibacterium prausnitzii between their habitual diet and EEN diet or the CD-TREAT diet.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult people
2. Normal weight (Body Mass Index: 18-25kg/m^2)
3. Stable weight the past month

Exclusion Criteria:

1. Acute or chronic illness (defined as illness which requires regular visits to health services)
2. Positive or negative energy balance (recent weight gain or loss, ±2 Kg the past month)
3. History of gut surgery
4. Use of antibiotics or steroids the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Gut Bacterial Composition | 12 months
  Gut microbiota composition measured by 16S rRNA gene amplicon sequencing, whole genome shotgun metagenomics and qPCR of selective bacterial species previously implicated in the onset of CD (e.g. Escherichia coli, Faecalibacterium prausnitzii, Bifidobacterium spp)
Gut Bacterial Metabolites | 12 months
  Gut microbiota metabolic activity as a measure of short chain fatty acids, hydrogen sulfide, lactate, ammonia and pH levels

SECONDARY OUTCOMES:
Dietary Intake | 12 months
  Dietary intake measured by a 7-day estimated dietary record

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Gerasimidis, BSc MSc PhD, Principal Investigator — University of Glasgow
Locations (1):
- School of Medicine, University of Glasgow / New Lister Building, Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svolos V, Hansen R, Nichols B, Quince C, Ijaz UZ, Papadopoulou RT, Edwards CA, Watson D, Alghamdi A, Brejnrod A, Ansalone C, Duncan H, Gervais L, Tayler R, Salmond J, Bolognini D, Klopfleisch R, Gaya DR, Milling S, Russell RK, Gerasimidis K. Treatment of Active Crohn's Disease With an Ordinary Food-based Diet That Replicates Exclusive Enteral Nutrition. Gastroenterology. 2019 Apr;156(5):1354-1367.e6. doi: 10.1053/j.gastro.2018.12.002. Epub 2018 Dec 11. PMID 30550821